CLINICAL TRIAL: NCT05512364
Title: Elacestrant for Treating ER+/HER2- Breast Cancer Patients With ctDNA Relapse
Brief Title: Elacestrant for Treating ER+/HER2- Breast Cancer Patients With ctDNA Relapse (TREAT ctDNA)
Acronym: TREAT ctDNA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Breast International Group (Other); Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-2129-BCG
Record Dates: First submitted 2022-08-22; First posted 2022-08-23 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: ER-positive Breast Cancer; HER2-negative Breast Cancer; Stage IIB Breast Cancer; Stage III Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — elacestrant; Tamoxifen; Letrozole; Anastrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): elacestrant 400 mg/day orally once daily on a continuous dosing schedule
  Interventions: Drug: Elacestrant
- Control arm (Active Comparator): standard endocrine treatment - the same they were receiving at the time of ctDNA detection
  Interventions: Drug: Tamoxifen; Drug: Letrozole 2.5mg; Drug: Anastrozole 1mg; Drug: Exemestane 25 MG

INTERVENTIONS:
Drug: Elacestrant — 400mg QD orally on a continuous dosing schedule
  Arms: Experimental arm
Drug: Tamoxifen — 20 mg QD orally on a continuous dosing schedule
  Arms: Control arm
Drug: Letrozole 2.5mg — 2.5 mg QD orally on a continuous dosing schedule
  Arms: Control arm
Drug: Anastrozole 1mg — 1 mg QD orally on a continuous dosing schedule
  Arms: Control arm
Drug: Exemestane 25 MG — 25 mg QD orally on a continuous dosing schedule
  Arms: Control arm

SUMMARY:
This is an international, multi-center, randomised, open label, superiority phase III trial of elacestrant vs standard endocrine therapy in patients with ER+/HER2- breast cancer and ctDNA relapse.

During the ctDNA screening phase, patients will be tested at different timepoints to detect the presence of ctDNA in their blood.

Patients who are found to be ctDNA-positive and have no evidence of distant metastasis, will be randomised 1:1 between standard endocrine treatment (the same they were receiving when tested ctDNA positive) versus elacestrant, provided they meet all eligibility criteria. After completion of the protocol treatment period, treatment will be left at the discretion of the treating physician.

DETAILED DESCRIPTION:
International, multi-center, randomised, open label, superiority phase III trial of elacestrant vs standard endocrine therapy in patients with ER+/HER2- breast cancer and ctDNA relapse.

1. ctDNA screening phase: After verification of the eligibility criteria for screening, patients will enter the ctDNA screening phase of the study in which plasma samples will be collected and tested with ctDNA assay to detect the presence of ctDNA. The test will be performed every 6 months from study entry until the end of accrual (approximately 5.7 years). During the screening phase, patients will be treated with standard adjuvant endocrine therapy [either tamoxifen or an aromatase inhibitor (exemestane, anastrozole or letrozole)] and followed-up as per standard of care. The outcome of the serial ctDNA assessments performed during the screening phase will be disclosed to investigators.

   Patients who are found to be ctDNA-negative at the end of the screening period will not be followed further in this study.

   Patients who are found to be ctDNA-positive at one of the screening time points will undergo an imaging work-up to assess the presence of distant metastases.

   Patients for whom the imaging work-up confirms no evidence of distant metastases or locoregional recurrence will be eligible for the randomised phase of the study provided they meet all other eligibility criteria. Patients for whom the imaging work-up shows evidence of distant metastases or locoregional recurrence will be excluded.
2. Randomised trial:

Patients will be randomised 1:1 within 4 weeks from the date of ctDNA detection (i.e., the date on which the results of the test are received) between standard endocrine treatment (the same they were receiving when tested ctDNA positive) versus elacestrant.

In the absence of a withdrawal criteria, treatment in both arms will be administered for:

* For patients on ET between 1 to 5 years (12 to 60 months) at the time of randomisation: 2 to 6 years (allowing for 7 years of ET at the end of the study treatment).
* For patients on ET between 5 to 7.5 years (60 to 90 months) at the time of randomisation: 2 years.

After completion of the protocol treatment period, treatment will be left at the discretion of the treating physician.

Patients in both arms will undergo intensive follow-up with ctDNA tests at week 4 and week 16 after randomisation and every 16 weeks thereafter for a maximum of 3 years (36 months or 156 weeks) to assess ctDNA kinetics. In addition, the occurrence of distant metastases, locoregional recurrences and second cancers will be assessed via yearly mammograms and bone scans and 16-weekly CT scans thorax/abdomen for a maximum of 3 years after randomisation. Afterwards, follow-up will continue as per standard of care. All randomised patients will be followed-up until 3 years after the enrolment of the last patient.

End of study:

End of study occurs when all the following criteria have been satisfied:

All patients have completed their end of study visit. If a patient discontinues the follow-up due to withdrawal of consent, loss to follow-up, or death, the end of study participation is defined as the time point when one of these events occurred The trial is mature for all analyses defined in the protocol and the database has been cleaned and frozen for these analyses.

ELIGIBILITY:
Inclusion Criteria:

1. ctDNA screening phase:

   Main inclusion criteria:

   • Female (both pre- and postmenopausal) or male patients with histologically confirmed ER positive (regardless of PR),

   HER2 negative breast cancer, according to local pathologist:
   * ER-positive defined as ≥ 10% of cells staining positive for ER or Allred proportion score ≥3
   * HER2-negative defined as a score of 0, 1+ by immunohistochemistry (IHC) or a negative in situ hybridization (ISH) based on single-probe average HER2 copy number, as per American Society of Clinical Oncology guidelines
   * Intermediate to high risk of recurrence after definitive treatment for early breast cancer, defined as:

   FOR PATIENTS TREATED WITH PRIMARY SURGERY:
   * Any patient with ≥ 4 positive axillary lymph nodes (stage pN2-3).
   * 1-3 positive axillary lymph nodes (stage pN1) and either:
   * Tumour size ≥ 5 cm or/and
   * Histologic grade 3 or/and
   * Ki67≥20% or/and
   * High genomic risk defined as Oncotype Dx Recurrence Score >=26, Mammaprint high risk, Prosigna score >40 or EPclin risk score >=4.0.
   * Negative axillary lymph nodes (stage pN0) and tumour size ≥ 5 cm and either
   * Histologic grade 3 a or/and
   * Ki67≥20% and/or
   * High genomic risk defined as Oncotype Dx Recurrence Score >=26, Mammaprint high risk, Prosigna score >60 or EPclin risk score >=4.0. FOR PATIENTS TREATED WITH NEOADJUVANT

   SYSTEMIC TREATMENT FOLLOWED BY SURGERY:
   * Patient may have received neoadjuvant endocrine therapy or neoadjuvant chemotherapy provided that:
   * The initial tumour and/or the tumour after surgery meet the criteria above defined for patients treated with primary surgery or the initial tumour was staged as cT4anyN and
   * There is no pathological complete response, defined as no invasive disease in the breast and axilla (ypT0/is ypN0).
   * Age ≥18 years
   * Patients must have received at least 1 year and up to 7.5 years of ET and planned to continue adjuvant ET during ctDNA screening phase
   * Previous adjuvant CDK4/6 inhibitor or PARP-inhibitor treatment is allowed provided it is completed
   * Invasive multicentric / multifocal disease is allowed provided that all the tested foci are ER+ HER2-. A sample from the highest-risk one, according to the investigator decision based on the size and grade, should be sent to Natera to build the patient ctDNA assay.
   * Available tumour sample from resected or biopsied tissue, with a tumour content of ≥20% (30% preferred) either before or after macro dissection (if performed) and a cell viability of a minimum 100 cells.
   * Core Needle Biopsies (CNB): recommended minimum of four (4) cores per block
   * Fine Needle Aspirates (FNA) are not accepted
   * The following sample types are acceptable:
   * 6-10 unstained slides (charged and unbaked) of 10μm each (or 12-19 unstained slides at 5 μm each), PLUS one contiguous H&E slide. Minimum total tissue thickness must be 60μm OR
   * FFPE tissue block with 25mm2 minimum surface area
   * Written informed consent must be given according to ICH/GCP, and national/local regulations.

   Main exclusion criteria:
   * Suspected recurrent disease or known conflicts with the inclusion and exclusion criteria for the randomised trial
   * Prior treatment with any SERD or investigational ER antagonist
   * Previous history of invasive breast cancer
   * Previous history of any other malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ.
   * Previous history of bone marrow and/or organ transplant
   * Bilateral breast cancer
   * Participation in another clinical study, with the exception of the SURVIVE study and observational (non-interventional) and non-drug intervention clinical studies. Note: patients participating in interventional studies may participate once they enter the follow-up period of the study
   * Blood transfusion within 3 months prior to registration or during the screening.
2. Randomised trial:

Main inclusion criteria:

* ctDNA positive according to the Signatera ctDNA assay (main study ctDNA test) or other ctDNA assay approved for diagnostic purposes.
* Patients must meet the eligibility criteria for the screening phase, with the exception of the tissue sample requirements.
* Patients must receive adjuvant ET at the time of the ctDNA positive test
* Absence of locoregional and/or metastatic disease and/or new malignancy, as investigated by:
* Mammogram (unilateral in case of mastectomy; not required in patients having undergone bilateral mastectomy) NOTE: if local investigator plans to use MRIs instead of mammograms during the study, MRI will have to be performed at baseline.
* CT thorax and abdomen/pelvis with IV contrast. In case of any contra-indications (medical or regulatory): CT thorax without contrast + MRI abdomen/pelvis.
* Technetium-99m bone scintigraphy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Adequate organ function
* Women of childbearing potential (WOCBP) must have a negative highly sensitive serum or urine pregnancy test within 7 days prior to randomisation.

Main exclusion criteria:

* Any unresolved toxic effect of prior therapies or surgical procedures of Grade ≥ 2 according to Common Terminology Criteria of Adverse Events (CTCAE) v5.0, with the exception of alopecia, peripheral neuropathy and other toxicities not considered a safety risk for the participant at investigator's discretion
* Unable or unwilling to avoid over-the-counter medications, dietary/herbal supplements, and/or foods that are moderate/strong inhibitors or inducers of CYP3A4 activity
* Known difficulty in tolerating oral medications or conditions which would impair absorption of oral medications
* Any of the following cardiovascular disorders within 3 months before enrolment:
* myocardial infarction
* stroke
* severe/unstable angina
* symptomatic cardiac arrhythmia
* prolonged QTcF ≥ Grade 3 (i.e., > 500 msec)
* heart failure ≥ Class III as defined by the New York Heart Association (NYHA) guidelines
* Child-Pugh Score greater than Class A
* Uncontrolled significant active infections (≥ grade 3 according to CTCAE version 5), including active hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency Virus (HIV)
* Coagulopathy or any history of coagulopathy within the past 6 months, including history of deep vein thrombosis or pulmonary embolism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2032-11-01 (Estimated); Study Completion 2035-11-01 (Estimated)

PRIMARY OUTCOMES:
Distant metastasis free survival (DMFS) | Final DFMS will be 6.25 years after the first patient randomised.
  Distant metastasis free survival (DMFS) defined as the time from randomisation until first distant metastatic recurrence or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
Invasive disease-free survival (iDFS) | Through study completion, up to 11.7 years
  According to the STEEP criteria, it's defined as the time between the date of randomisation and the date of the first occurrence of one of the following events: loco-regional disease recurrence, distant metastasis, invasive contralateral breast cancer, invasive non-breast second cancer, or date of death from any cause
Relapse-free survival (RFS) | Through study completion, up to 11.7 years
  Relapse-free survival (RFS) rate according to the STEEP criteria, including locoregional recurrence, distant metastasis, deaths from any cause as events
Overall survival rate | Through study completion, up to 11.7 years
  Overall survival rate
  • Safety including but not limited to all adverse events, serious adverse events, laboratory abnormalities graded according to CTCAE version 5.0
Adverse events | as of randomization until 30 days after administration of the last dose of protocol treatment.
  Safety including but not limited to all adverse events, serious adverse events, laboratory abnormalities graded according to CTCAE version 5.0
Health Related Quality of Life QLQ-C30 | weeks 4, 16, 32, 48, 64 and 80
  European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core-30 (QLQ-C30). This is a patient-reported questionnaire composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. All of the scales and single-item measures range in score from 0 to 100.A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
  Assessments will be performed at 21 days before randomisation, 4 weeks, 16 weeks, 32 weeks, 48 weeks, 64 weeks, and 80 weeks after randomisation using the following measures: QLQ-C30
Health Related Quality of Life EORTC IL146 | weeks 4, 16, 32, 48, 64 and 80
  Health-related quality of life (HRQoL) is a secondary endpoint in this trial. HRQoL assessment aims at
  1. establishing the patient-reported tolerability profile in each treatment arm.
  2. comparing the patient-reported benefit between the two treatment arms.
  Assessments will be performed at 21 days before randomisation, 4 weeks, 16 weeks, 32 weeks, 48 weeks, 64 weeks, and 80 weeks after randomisation using the following measures: EORTC IL146.
Health Related Quality of Life QLQ-BR42 | weeks 4, 16, 32, 48, 64 and 80
  Health-related quality of life (HRQoL) is a secondary endpoint in this trial. HRQoL assessment aims at
  1. establishing the patient-reported tolerability profile in each treatment arm.
  2. comparing the patient-reported benefit between the two treatment arms.
  Assessments will be performed at 21 days before randomisation, 4 weeks, 16 weeks, 32 weeks, 48 weeks, 64 weeks, and 80 weeksafter randomisation using the following measures:QLQ-BR42

CONTACTS AND LOCATIONS:
Overall Officials: Michail Ignatiadis, Study Chair — Institut Jules Bordet, Belgium; Emmanouil Saloustros, Study Chair — General University Hospital of Larissa, Greece
Locations (94):
- Belgium (11):
  - Institut Jules Bordet, Anderlecht
  - AZ KLINA, Brasschaat
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hopital de Charleroi - Site Notre Dame, Charleroi
  - CHU Helora Pole Hospitalier Jolimont - Hopital Jolimont, Haine-Saint-Paul
  - AZ Groeninge Kortrijk - Campus Kennedylaan, Kortrijk
  - U.Z. Leuven - Campus Gasthuisberg, Leuven
  - CHU Site Sainte-Elisabeth-UCL Namur, Namur
  - AZ Delta - Campus Rumbeke, Roeselare
  - AZ Turnhout - Campus Sint Elisabeth, Turnhout
  - Centre Hospitalier Regional Verviers, Verviers
- Cyprus (2):
  - German Oncology Center, Limassol
  - Bank Of Cyprus Oncology Centre, Stróvolos
- France (13):
  - CH de La Cote Basque - Saint Leon, Bayonne
  - Clinique Belharra-Ramsay Sante, Bayonne
  - Centre de Radiotherapie Pierre Curie, Beuvry
  - Centre Hospitalier - Boulogne Sur Mer, Boulogne-sur-Mer
  - CHU de Lyon - Hopital Femme Mere Enfant, Bron
  - Societe de Recherche Oncologique Clinique 37, Chambray-lès-Tours
  - Hopital de Douai- Centre Leonard de Vinci, Dechy
  - CHU de Limoges - Hopital Dupuytren, Limoges
  - CHU de Lyon - Hopital De La Croix Rousse, Lyon
  - Polyclinique De Gentilly - Centre d'Oncologie, Nancy
  - CHU de Lyon - Hopital Lyon Sud, Pierre-Bénite
  - Institut Curie - l'Hopital de St Cloud, Saint-Cloud
  - CHU de Toulouse - Institut Claudius Regaud - IUCT oncopole, Toulouse
- Germany (17):
  - Universitaetsklinikum Aachen AOR - Medizinische Fakultaet der RWTH, Aachen
  - Gemeinschaftspraxis Augsburg, Augsburg
  - Evangelisches Krankenhaus -Bergisch Gladbach, Bergisch Gladbach
  - Marienhospital Bottrop gGmbH, Bottrop
  - Hamatologische Onkologische Praxis Im Medicum, Bremen
  - St Elisabeth-Krankenhaus, Cologne
  - Universitaetsklinikum Carl Gustav Carus (TUD), Dresden
  - Medizinische Hochschule Hannover, Hanover
  - Gemeinschaftspraxis Dr. Pourfard / Dr. Uleer, Hildesheim
  - Klinikum Kassel Gmbh, Kassel
  - MVM MbH -Onkologie UnterEms, Leer-Papenburg-Emden, Leer
  - Busch MCZ GmbH, Mühlhausen
  - Klinikum Nuernberg- Standort Nord, Nuremberg
  - Klinikum Ernst von Bergmann gemeinnützige GmbH, Potsdam
  - Universitaetsklinikum Tuebingen-calwerstrasse, Tübingen
  - Universitaetsklinikum Ulm-Michelsberg, Ulm
  - HELIOS Kliniken - Helios Klinikum Wuppertal - Klin. Univ. Witten / Herdecke, Wuppertal
- Greece (2):
  - Diagnostic & Therapeutic Center of Athens Hygeia Hospital S.A., Athens
  - General University Hospital of Larissa, Larissa
- Ireland (3):
  - Mater Private Hospital, Dublin
  - St. James'S Hospital, Dublin
  - Beacon Hospital, Dublin
- Italy (16):
  - Centro Di Riferimento Oncologico, Aviano
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Univ. of Florence -Azienda Ospedaliero-Universitaria Careggi, Florence
  - IRCCS Azienda Policlinico San Martino, Genova
  - Azienda USL IRCCS Di Reggio Emilia Guastalla, Guastalla
  - Ospedale Alessandro Manzoni, Lecco
  - Azienda Unita Locale Socio-Sanitaria N. 9-Mater Salutis Hospital, Legnano
  - IRCCS Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola
  - University Hospital of Cagliari Duilio Casula Hospital Unit (Policlinico), Monserrato
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Istituti Clinici Scientifici Maugeri, Pavia
  - San Maria della Misericordia Hospital, Perugia
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Azienda USL IRCCS Di Reggio Emilia - Maria Nuova, Reggio Emilia
  - AUSL Romagna - AUSL Della Romagna - Infermi Hospital -Rimini, Rimini
- Netherlands (7):
  - Flevoziekenhuis Stichting, Almere Stad
  - Amsterdam UMC - locatie VUMC, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Haaglanden Medisch Centrum, Leidschendam
  - Ikazia Ziekenhuis, Rotterdam
  - Sint Antonius - St Antonius Ziekenhuis Utrecht, Utrecht
  - VieCuri - Medisch Centrum voor Noord-Limburg - Locatie Venlo, Venlo
- Spain (19):
  - Hospital General Universitario Doctor Balmis, Alicante
  - Hospital Universitario De Cruces, Barakaldo
  - Hospital Clinico Universitario - Virgen De La Arrixaca, El Palmar
  - ICO Girona - Hospital Doctor Josep Trueta, Girona
  - Hospital Universitario Virgen De Las Nieves, Granada
  - Hospital Universitario Clinico San Cecilio, Granada
  - ICO L'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital Universitari Arnau De Vilanova, Lleida
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospitales HM Sanchinarro-CIOCC, Madrid
  - Althaia Xarxa Assistencial Universitaria De Manresa Fundacio Privada, Manresa
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario de Navarra, Pamplona
  - Hospital Sant Joan de Reus, Reus
  - Hospital Quironsalud Sagrado Corazon, Seville
  - University Hospital Virgen del Rocio, Seville
  - Hospital Universitario Virgen De La Macarena, Seville
  - Hospital Clinico Universitario De Valencia, Valencia
  - Hospital Universitario Y Politecnico La Fe, Valencia
- Sweden (2):
  - Sodra Alvsborgs Sjukhus - Vastra Gotalandsregionen, Borås
  - Karolinska University Hospital, location Solna, Stockholm
- Switzerland (2):
  - Kantonsspital Frauenfeld- Breast Unit Thurgau, Frauenfeld
  - Buergerspital Solothurn -Brustzentrum, Solothurn

IPD SHARING:
Plan to Share IPD: No